CLINICAL TRIAL: NCT01931384
Title: A Randomized Controlled Comparison of Human Chorionic Gonadotrophin as Luteal Phase Support in Frozen-thawed Embryo Transfer Cycles
Brief Title: A Study of Human Chorionic Gonadotrophin as Luteal Phase Support in Frozen Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU-VL-LPSRCT
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Subfertility
Keywords: Luteal phase support; Human chorionic gonadotrophin; frozen-thawed embryo transfer cycle
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): luteal phase support using Human chorionic gonadotrophin 1500 IU intramuscular injection will be given on the day of FET and 6 days later.
  Interventions: Drug: Human chorionic gonadotrophin
- control group (Placebo Comparator): normal saline (placebo) intramuscular injection will be given on the day of FET and 6 days later
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human chorionic gonadotrophin — luteal phase support using Human chorionic gonadotrophin 1500 IU intramuscular injection will be given on the day of FET and 6 days later.
  Arms: Intervention group
Drug: Placebo — Normal saline intramuscularly on the day of embryo transfer and 5 days after embryo transfer.
  Other Names: Normal saline
  Arms: control group

SUMMARY:
A randomised trial on the use of luteal phase support in frozen-thawed embryo transfer cycles.

The hypothesis of the study is that the use of luteal phase support with human chorionic gonadotrophin would increase the pregnancy rate in frozen-thawed embryo transfer cycles.

DETAILED DESCRIPTION:
Trial design:

-A total of 450 women undergoing FET in the Centre of Assisted Reproduction and Embryology, The University of Hong Kong-Queen Mary Hospital, will be recruited. They will be randomized into one of the following two groups by computer-generated random numbers:

Group I: luteal phase support using HCG 1500 IU intramuscular injection will be given on the day of FET and 6 days later.

Group II: normal saline (placebo) intramuscular injection will be given on the day of FET and 6 days later.

Treatment:

Ovarian stimulation protocol:

All women received ovarian stimulation according to the standard protocol of the Centre. HCG is given intramuscularly when the leading follicle reaches 18 mm in mean diameter. Oocyte retrieval is carried out 36 hours after the HCG trigger. A maximum of two embryos will transferred and any excess good quality embryos will be frozen two days after the retrieval.

FET cycle:

FET is carried out at least 2 month after the stimulated cycle if the patient fails to get pregnant in the stimulated IVF cycle and there is at least one frozen embryo. Frozen embryos after thawing are transferred in natural cycles for those women having regular ovulatory cycles, during which the patient is monitored daily for serum estradiol ad luteinising hormone levels from 18 days before the expected date of the next period.

The transfer is performed by the team clinician on the third day after the luteinising hormone surge and a maximum of two normally cleaving embryos are replaced according to our standard protocol. The luteal phase is supported as per randomization arm. Before the embryo transfer, the patient is interviewed by a designated research nurse who will explain the purpose of this study. Patients consenting to take part in the study will be assigned into one of the two study arms specified in an opaque envelope according to a computer-generated randomization list. The envelope will be read and injection (HCG or placebo as normal saline) given by a service nurse not involved in the study. Blood will be taken on day 6 after FET before the patient receives the second dose of HCG or placebo. A urine pregnancy test will be performed 16 days after the FET. In case of pregnancy, the outcome of pregnancy will be traced afterwards and used for analysis. Luteal phase support is not continued in those who get pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Normal uterine cavity shown on pelvic scanning during the stimulated IVF cycle
* Endometrial thickness >=8mm in FET cycles

Exclusion Criteria:

* Subjects requiring clomid-induced cycles and hormonal replacement (HRT) cycles
* History of previous FET cycles within the study period
* Blastocyst transfer
* Use of donor oocytes
* Presence of hydrosalpinx not corrected surgically prior to FET
* Refusal to join the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 4 months
  ongoing pregnancy rate which is defined as the number of on-going pregnancies beyond 10-12 weeks gestation per transfer cycle

SECONDARY OUTCOMES:
Rate of pregnancy loss per number of transfer cycles | 4 months
  The pregnancy loss after embryo transfer counted

OTHER OUTCOMES:
Implantation rate | 4 months
  number of gestational sacs per number of embryos transferred
Hormonal profile | 2 weeks
  Hormonal profile including the serum oestradiol, progesterone and hCG concentrations at the mid-luteal phase (day 6 after FET)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Chi Yan Lee, MBBS, Principal Investigator — HKU / QMH
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lee VCY, Li RHW, Yeung WSB, Pak Chung HO, Ng EHY. A randomized double-blinded controlled trial of hCG as luteal phase support in natural cycle frozen embryo transfer. Hum Reprod. 2017 May 1;32(5):1130-1137. doi: 10.1093/humrep/dex049. PMID 28333292